CLINICAL TRIAL: NCT06297239
Title: Argentine Registry for the Study of Lipoprotein a
Brief Title: Argentine Registry of Lp(a)
Acronym: GAELpa
Status: Recruiting | Type: Observational
Sponsor: School of Medicine. National University of Cuyo (Other)
Responsible Party: Sponsor
Other Study IDs: UC001
Record Dates: First submitted 2024-02-27; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Lp(A); Hypercholesterolemia; Cardiovascular Diseases; Diabete Type 2; Hypertension
Keywords: LP(a); Cardiovascular risk
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Argentine Registry on Lipoprotein(a) (LP(a)), orchestrated by the Argentine Group for LP(a) Study, stands as a pioneering and extensive prospective initiative. This registry systematically collects geolocation data, including patient postal codes, demographic information, and a multifaceted array of health parameters to unravel the intricate associations surrounding LP(a) levels.

The dataset encompasses diverse patient characteristics, ranging from standard metrics like blood pressure, weight, and race to broader factors such as diabetes, smoking habits, menopausal status, and hypothyroidism. This holistic approach enables a nuanced exploration of the interplay between LP(a) levels and various risk factors, providing invaluable insights for both clinical and public health considerations.

One distinctive feature of this registry lies in its focus on medication history, shedding light on the impact of routine pharmaceutical interventions on LP(a) profiles. Additionally, it delves into the intricate web of inflammatory diseases, recognizing their potential role in LP(a) modulation.

Genetic predispositions are meticulously examined, with a specific emphasis on identifying homozygous and heterozygous variants associated with hypercholesterolemia. This genetic dimension adds a layer of complexity to the understanding of LP(a) dynamics, contributing significantly to the ongoing discourse on cardiovascular risk.

The prospective nature of this registry allows for dynamic analyses, fostering a continuous exploration of emerging patterns and trends. By amalgamating geographical, clinical, and genetic data, the Argentine LP(a) Registry emerges as a comprehensive platform poised to unlock novel facets of LP(a) biology and its implications for cardiovascular health. As the dataset matures, it holds the promise of guiding personalized interventions and refining risk stratification strategies, thereby advancing the landscape of preventive cardiovascular care.

ELIGIBILITY:
Inclusion Criteria: Adult patients with validated Lp(a) values -

Exclusion Criteria: Associated pathologies that can increase the Lp(a) value in a non-specific manner

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult patients residing in Argentina
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of high level of Lp(a) | 2 years
  prevalence of high level of Lp(a)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Corral, MD, Study Chair — FASTA University
Locations (1):
- Universidad Nacional de Cuyo, Mendoza, Argentina